CLINICAL TRIAL: NCT02413151
Title: Exercise Training Following Cardiac Resynchronization Therapy in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Maria Helena Santa-Clara Pombo Rodrigues, Assistant Professor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTDC/DES/120249/2010
Record Dates: First submitted 2015-03-25; First posted 2015-04-09 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Resynchronization Therapy; Chronic Heart Failure
Keywords: Exercise training; Cardiac resynchronization therapy; Autonomic nervous system modulation; Chronic Heart failure
MeSH Terms: interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Training Program (Experimental): The exercise sessions will be hospital-based, 3 times a week for 60 minutes each, on non-consecutive days for 6 months. Selected the aerobic interval training (AIT) method for the development of cardiopulmonary system and the inclusion of resistance and sensorimotores exercises. The AIT comprises 4 interval training periods (high intensity) and 3 active pauses (moderate intensity) between interval training periods.
  Interventions: Behavioral: Exercise training program; Device: Cardiac resynchronization therapy (CRT)
- Control (Active Comparator): Regular lifestyle
  Interventions: Device: Cardiac resynchronization therapy (CRT)

INTERVENTIONS:
Behavioral: Exercise training program — The exercise sessions will be hospital-based, 3 times a week for 60 minutes each, on non-consecutive days for 6 months. Selected the aerobic interval training (AIT) method for the development of cardiopulmonary system and the inclusion of resistance and sensorimotores exercises. The AIT comprises 4 interval training periods (high intensity) and 3 active pauses (moderate intensity) between interval training periods. The patient will warmup for 10 minutes at 50% to 60% of HRpeak from CPET, before walking to four 4 minutes intervals at 90 to 95% of peak HR. Each interval, including the last one, is separate by 3 minutes active pauses, walking at 60% to 70% of HRpeak. Total aerobic exercise time at this moment will be 28 minutes and will be maintain to the end of ExT intervention period.
  Arms: Exercise Training Program
Device: Cardiac resynchronization therapy (CRT) — Implantation will be performed according to standard techniques of biventricular pacing. The CRT includes a generator and three leads, used to correct ventricular dyssynchrony.

SUMMARY:
Cardiac resynchronization therapy(CRT) is recommended to reduce mortality and morbidity in chronic heart failure(CHF) patients New York Heart Association(NYHA) class III-IV who are symptomatic despite optimal medical therapy, with a reduced left ventricular(LV) ejection fraction(LVEF) and prolonged complex QRS. CRT improves the prognosis however, despite the improvement, all major trials have demonstrated that one third of the patients are non-responders to CRT. Three months after the CRT implant, the responders have a significant increase in endothelial function(EntF), a decrease in the LV end-systolic volume, and increase in LVEF, 6 minute walk test(6MWT), improvements in NYHA class and quality of life. It is currently unknown if adding an exercise training(ExT) program following CRT provides better clinical outcomes than CRT alone. Prior studies on CRT and ExT have been preliminary in nature, but suggest small improvements in functional capacity(FC). The correction of endothelial dysfunction is associated with a significant improvement in exercise capacity evidenced by a 26%increase in peak oxygen uptake. These findings are important because CHF patients with the greatest sympathetic activation and the most reduced EntF have the poorest prognosis. Our experience with coronary artery disease patients, and most recently data in patients with CHF show that an ExT program that combines aerobic exercise(AE) and resistance exercise training are more effective than an AE program alone, and the aerobic interval training showed better improvements than continuous endurance training. It is unknown how CHF with more severe functional limitations responds to ExT and, more important, the explanation of the physiological mechanism that can explain the improvements as a consequence of ExT. This lack of scientific information is urgent since this is the group of patients that normally is targeted for CRT. The investigators propose to use a stratified randomized longitudinal study to determine the additional effects of a 6 month ExT in addition to CRT in NYHA stage III-IV HF patients. The aims of the study are:1-to determine whether a long-term ExT program follow the CRT provides better clinical outcomes than CRT alone and 2-To identify the mechanisms of the hypothesize improvement. The results of this project will represent an important contribution by understanding the role of ExT after CRT NYHA stage III-IV heart failure(HF) patients, an understudied population with poor clinical outcome. Understanding the potential mechanisms associated with clinical improvement and outcome is essential for the rehabilitative process to develop new innovative therapies in this high risk population. The investigators will use state-of-art methods including an integrated assessment autonomic nervous system(ANS) and arterial function using 123I-MIBG scintigraphy.

DETAILED DESCRIPTION:
Literature Review Generally CHF patients have reduced exercise capacity, with main symptoms of effort intolerance, early fatigue and breathlessness.They also exhibit increased peripheral and central chemosensitivity, impaired sympathovagal balance with sympathetic activity (SA) predominance, and depressed baroreflex n control. Compared with myocardium of healthy controls, the myocardium of patients with chronic LV dysfunction is characterized by a significant reduction of pre-synaptic norepinephrine (NE) uptake and post-synaptic beta adrenoceptor density.There is generalized increased SA in the heart of patients with CHF that might contribute to the remodeling process of the LV. This concept is consistent with the finding that down-regulation of myocardial beta-adrenoceptor density, measured using positron emission tomography with 11C-CGP-12177, soon after acute myocardial infarction (MI) is predictive of the occurrence of LV dilatation at follow-up. Myocardial beta-adrenoceptor density appears reduced in patients with HF due to dilated cardiomyopathy and down-regulation of myocardial beta-adrenoceptor is more pronounced in patients with hypertrophic cardiomyopathy who proceed to LV dilation and HF. Therefore, myocardial beta-adrenoceptor down-regulation may be a general nonspecific response to stress and could be due to a locally increased amount of NE in the synaptic cleft. The sustained hyperactivity of the SA observed in HF is the consequence of several mechanisms including increased central sympathetic outflow, altered neuronal NE reuptake, and facilitation of cardiovascular response to sympathetic stimulation by angiotensin II. CRT is an accepted treatment for patients with moderate-to-severe CHF and intraventricular conduction delay. Intraventricular conduction delays, identified by a QRS interval of 120 msec or more on a 12-lead electrocardiogram (ECG), occur in up to a third of patients with severe systolic HF and are associated with dyssynchronous contraction of the LV, leading to impaired emptying and, in some patients, mitral regurgitation. Abnormal atrioventricular coupling (identified by a prolonged PR interval) and interventricular dyssynchrony, identified on an echocardiogram, may also occur. CRT with atrialsynchronized biventricular pacing often improves cardiac performance immediately, by increasing stroke volume (SV) and reducing mitral regurgitation. Randomized trials involving patients with severe HF showed that CRT resulted in a reduction in symptoms and improved FC, a reduction in the number of hospitalizations for worsening HF, and increased survival. ExT in CHF produce meaningful improvements in peak oxygen consumption (VO2peak) with an expected average improvement of 17%. This is particularly important since improvement in FC is related to the improvement in neurohormonal activation, peripheral abnormalities and ventilatory function. Submaximal exercise capacity (SubMaxExC) is also improved, as assessed by a significant increase in the ventilatory anaerobic threshold (VAT) and in 6-MWT. The improvement in SubMaxExC of CHF patients (NYHA II-III) was probably due to peripheral training adaptations in skeletal muscle mass (SMM). Theoretically, by improving SMM strength, a lower % of maximal contraction would be used to do a similar amount of work following training. A lower relative muscle contraction would be expected to produce less blood lactate, thereby decreasing the need for carbon dioxide (CO2) elimination, thus increasing the VAT. The improvement in VAT is important as it would allows patients to exercise longer and harder without negative alterations in ventricular dynamics associated with the VAT and could possibly delay the onset of the ischemic threshold. To severe CHF patients, the truly meaning of improvement SubMaxExC as effect of ExT is related to QOL since the engagement in daily activities does not demand VO2peak. All the previous studies were done with low to moderate risk patients but high risk patients probably have a greater need in order to lead a normal, independent life. Results from previous studies with CHF showed that ExT reduces NE levels at rest and during exercise, decreases central sympathetic nerve outflow as measured by microneurography. ExT also enhances vagal control with a shift away from sympathetic activity, and improves heart rate (HR) variability and HR recovery with a return to a better sympathetic-vagal balance. Moreover, ExT produces significant reduction in the local expression of cytokines such as interleukin (IL)-6 and inducible nitric oxide synthase (iNOS) in the SMM of CHF patients and has a beneficial effect on peripheral inflammatory markers reflecting monocyte/macrophage-endothelial cell interaction. These local anti inflammatory effects of ExT may attenuate the catabolic wasting process associated with the progression of CHF. This can be an important issue since inflammatory responses plays a pathogenic role in the development and progression of CHF. Probably the impaired availability of nitric oxide (NO) is responsible for the impaired endothelium dependent relaxation of peripheral resistance and conduit arteries and may contribute to the reduced FC in CHF and other severe symptoms. Also endothelium-independent vasodilatation abnormalities may relate to a combination of impaired smooth muscle responsiveness to NO, impaired of NO diffusion to the smooth muscle or structural alterations in arterial compliance associated with CHF. The combination of ExT in CRT is not been well-investigated. One small-scale pilot study (not randomized ) suggested that functional capacity improved. More recently, Patwala et al. reported improvements in quality of life (QOL) and VO2peak through improved SMM performance with the addition of a 3-month ExT 3-month after the CRT. In this study, all the patients were in class III of NYHA and an ExT only 3 months in duration. Little is known about ExT for elderly severe CHF patients.

Plan and Methods The purpose of this research project is to determine the effects of adding ExT to CRT on clinical status, ANS function, in ischemic and nonischemic cardiomyopathy patients with moderate to severe CHF. The investigators will evaluate the following specific aims: 1- To determine the effects of a long-term ExT program following CRT provides on clinical outcome; 2-Identify the mechanisms of the hypothesized improvements in clinical status. The primary end points for aim 1 are the clinical status, namely NYHA functional class, all-cause mortality, hospitalization rate, cardiac function and maximal and SubMax FC. For aim 2 the SA, HRV, HRR and blood endothelin-1, brain natriuretic peptide (BNP), IL-6, tumor necrosis factor (TNF)-a and C reactive protein (CRP). As secondary end points the investigators will analyze neuromuscular function(NMF), body composition(BC) and QOL. Relevance: Due to increased prevalence of CHF and consequent implications for mortality and morbidity rates, the prognosis of HF has improved in the past 20 years, but it remains a serious condition with a markedly increased risk of death in the early period after onset of the syndrome. In population studies, there is 10% mortality by 30 days. For those who survive this early high-risk period, the 5-year mortality is 54% in men and 40% in women. In clinical trials of CHF therapy, 50% of deaths are due to sudden death and progressive HF accounts for around 30% of deaths, this latter proportion increasing as symptomatic severity increases.In population studies including patients with new-onset HF, progressive HF appears to be the single most common cause of death (52%), with sudden death accounting for only 22% of deaths within the first 6 months of diagnosis.ExT has been shown to be effective in CHF patients NYHA II-III, as it improves autonomic control by enhancing vagal tone and reducing sympathetic activation, improves exercise FC, QOL, SMM, vasodilator capacity, endothelial dysfunction and decrease oxidative stress, hospitalization and mortality%. No information is available in more severe patients and they are the patients that are in most need and their treatment will also significantly impact heath care costs. Moreover, scientific research is absent on the effects of ExT after CRT on severe CHF patients and there is no information on the effects of both therapies on ANS. Thus, the proposed project will address a number of important gaps in scientific knowledge with potentially large clinical benefits. Methods: The investigators will use a controlled stratified experimental design, using a longitudinal approach with 3 assessment time points: baseline, before the cardiac implant (CI) (M1); at 3 (M2) and 6-month (M3) after the experimental therapy (ET). It will be a continuum of recruitment during the 24 month but the study protocol it will be the same for all patients. The study will employ state of the art methods for ANS analysis, namely the Scintigraphy with 123I-meta-iodobenzylguanidine (123I-MIBG). The investigators will evaluate both clinical, physiological and QOL outcomes. The assessment of cardiac sympathetic neuronal activity with 123I-MIBG, a radio-labelled analogue of NE, will improve the understanding of the mechanisms responsible for increased sympathetic activity in HF, and how sympathetic overactivity exerts its deleterious actions. This technique offers a huge advantage in order to understand what happens in the heart, compared to the more commonly used technique of Muscle Sympathetic Nerve Activity. The inclusion of a M2 assessment will allow us to update the exercise intensity and also to conduct initial data analysis. Also the technique chosen in our project for group assignment (stratified by age and etiology randomization), provides the best opportunity to evaluate if the expected changes will be related with ET since patients with different age and etiology responded differently to ExT. The ExT design was done based on Wisloff's results. The AE will be developed with an AIT since previous results showed better results but due to the clinical status of our patients and longer intervention duration we will employ a different (slower) exercise prescription progression. We will begin with shorter aerobic intervals and only at the end of the 2nd month the investigators will use the same protocol as Wisloff et al. Compared with continuous exercise training methods, this method allows patients with HF to complete short periods of exercise at high intensity (which stress the heart's ability) but without deleterious effects of undue stress and fatigue. Another difference in the ExT program is the incorporation of resistive and sensoriomotor exercises (SME). These types of exercises will improve the lack of SMM of the CHF patients producing positive consequences in activities of daily life and QOL, and will enhance muscle performance of muscles not involved in the aerobic mode of exercise. This project can provide evidence for a useful and powerful treatment to reduce the high sympathetic activation (SA) that leads to an endothelial dysfunction contributing to both central and peripheral impairments in patients with severe CHF. In CHF patients, SA is initially increased as a compensatory mechanism; however, chronically elevated stimulation of the adrenergic system is associated with sustaining the process of myocardial remodeling. Another consequence is endothelial dysfunction manifested as impaired endothelium-dependent relaxation of peripheral resistance and conduit arteries, most probably due to impaired availability of NO. Besides the expected changes from the CRT we hypothesize that adding an ExT protocol that use the AIT and inclusion of endurance and SME to these patients will maximize both clinical and physiological outcomes. Our project will be the first to provide evidence for sympathetic and parasympathetic ANS action on the heart itself, and how these may be altered over 6 month of ET in patients with severe CHF. The combination of the selected assessment techniques will allow an overview of the expected adaptations and the underlying mechanisms. To our knowledge this project will be the first to address with precise and valid methods the benefits of a 6- month ExT program just after CRT on the ANS of moderate-to-severe CHF patients. Linking these results with NMF, BC, QOF and clinical status improvements will contribute to further understand the impact of ExT on overall health status of these patients. Also, the longer period of the ExT program and the inclusion of the M2 assessment will allow a more accurate analysis of the change process. Expected results: This study will firstly contribute to a better understanding of the implications of a combined therapy in CHF patients. This study can provide an extensive characterization of changes in ANS both central and peripheral, which will be of great value for stabilization or regression of the disease with direct impact in patient's daily life. It is expected that the ExT group compared with the control group will improve all the physiological variables included in the project as was observed in previous studies with less severe CHF patients and this will lead to improvements in clinical status. The investigators also expect that ExT group show a better improvement in the clinical outcomes and in health related QOL leading to a decrease in overall health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure (CHF), classified in NYHA functional class III or IV;
* Receiving optimal medical therapy for CHF (including an angiotensin-converting enzyme inhibitor or an angiotensin receptor blocker and a beta-blocker unless a contraindication is evident) with a stable condition for more than 1 month (no hospitalization for HF, no change in medication, and no change in NYHA functional class);
* Left ventricular ejection fraction (LVEF) < 35%;
* QRS duration ≥ 120 ms.

Exclusion Criteria:

* If they are younger than 18 years or are unable to sign informed consent;
* Patients who had been treated with an intravenous inotropic agent within the 30 days prior to implantation (these medications affect endothelial function after they are discontinued);
* Unstable angina pectoris;
* Orthopedic or neurological limitations to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helena Santa-Clara Pombo Rodrigues, PhD, Principal Investigator — University of Lisbon
Locations (1):
- Santa Marta Hospital, Lisbon, Portugal

REFERENCES:
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Bax JJ, Abraham T, Barold SS, Breithardt OA, Fung JW, Garrigue S, Gorcsan J 3rd, Hayes DL, Kass DA, Knuuti J, Leclercq C, Linde C, Mark DB, Monaghan MJ, Nihoyannopoulos P, Schalij MJ, Stellbrink C, Yu CM. Cardiac resynchronization therapy: Part 1--issues before device implantation. J Am Coll Cardiol. 2005 Dec 20;46(12):2153-67. doi: 10.1016/j.jacc.2005.09.019. PMID 16360042
- [Background] Akar JG, Al-Chekakie MO, Fugate T, Moran L, Froloshki B, Varma N, Santucci P, Wilber DJ, Matsumura ME. Endothelial dysfunction in heart failure identifies responders to cardiac resynchronization therapy. Heart Rhythm. 2008 Sep;5(9):1229-35. doi: 10.1016/j.hrthm.2008.05.027. Epub 2008 Jul 23. PMID 18774094
- [Background] Patwala AY, Woods PR, Sharp L, Goldspink DF, Tan LB, Wright DJ. Maximizing patient benefit from cardiac resynchronization therapy with the addition of structured exercise training: a randomized controlled study. J Am Coll Cardiol. 2009 Jun 23;53(25):2332-9. doi: 10.1016/j.jacc.2009.02.063. PMID 19539142
- [Background] Tabet JY, Meurin P, Driss AB, Weber H, Renaud N, Grosdemouge A, Beauvais F, Cohen-Solal A. Benefits of exercise training in chronic heart failure. Arch Cardiovasc Dis. 2009 Oct;102(10):721-30. doi: 10.1016/j.acvd.2009.05.011. Epub 2009 Sep 15. PMID 19913773
- [Background] Hambrecht R, Fiehn E, Weigl C, Gielen S, Hamann C, Kaiser R, Yu J, Adams V, Niebauer J, Schuler G. Regular physical exercise corrects endothelial dysfunction and improves exercise capacity in patients with chronic heart failure. Circulation. 1998 Dec 15;98(24):2709-15. doi: 10.1161/01.cir.98.24.2709. PMID 9851957
- [Background] Santa-Clara H, Fernhall B, Baptista F, Mendes M, Bettencourt Sardinha L. Effect of a one-year combined exercise training program on body composition in men with coronary artery disease. Metabolism. 2003 Nov;52(11):1413-7. doi: 10.1016/s0026-0495(03)00320-2. PMID 14624399
- [Background] Santa-Clara H, Fernhall B, Mendes M, Sardinha LB. Effect of a 1 year combined aerobic- and weight-training exercise programme on aerobic capacity and ventilatory threshold in patients suffering from coronary artery disease. Eur J Appl Physiol. 2002 Oct;87(6):568-75. doi: 10.1007/s00421-002-0675-4. Epub 2002 Jul 30. PMID 12355198
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] Caldwell JH, Link JM, Levy WC, Poole JE, Stratton JR. Evidence for pre- to postsynaptic mismatch of the cardiac sympathetic nervous system in ischemic congestive heart failure. J Nucl Med. 2008 Feb;49(2):234-41. doi: 10.2967/jnumed.107.044339. Epub 2008 Jan 16. PMID 18199620
- [Background] Spyrou N, Rosen SD, Fath-Ordoubadi F, Jagathesan R, Foale R, Kooner JS, Camici PG. Myocardial beta-adrenoceptor density one month after acute myocardial infarction predicts left ventricular volumes at six months. J Am Coll Cardiol. 2002 Oct 2;40(7):1216-24. doi: 10.1016/s0735-1097(02)02162-9. PMID 12383568
- [Background] Merlet P, Delforge J, Syrota A, Angevin E, Maziere B, Crouzel C, Valette H, Loisance D, Castaigne A, Rande JL. Positron emission tomography with 11C CGP-12177 to assess beta-adrenergic receptor concentration in idiopathic dilated cardiomyopathy. Circulation. 1993 Apr;87(4):1169-78. doi: 10.1161/01.cir.87.4.1169. PMID 8096441
- [Background] Choudhury L, Rosen SD, Lefroy DC, Nihoyannopoulos P, Oakley CM, Camici PG. Myocardial beta adrenoceptor density in primary and secondary left ventricular hypertrophy. Eur Heart J. 1996 Nov;17(11):1703-9. doi: 10.1093/oxfordjournals.eurheartj.a014754. PMID 8922919
- [Background] Middlekauff HR. How does cardiac resynchronization therapy improve exercise capacity in chronic heart failure? J Card Fail. 2005 Sep;11(7):534-41. doi: 10.1016/j.cardfail.2005.03.002. PMID 16198250
- [Background] Smart N, Marwick TH. Exercise training for patients with heart failure: a systematic review of factors that improve mortality and morbidity. Am J Med. 2004 May 15;116(10):693-706. doi: 10.1016/j.amjmed.2003.11.033. PMID 15121496
- [Background] Hambrecht R, Gielen S, Linke A, Fiehn E, Yu J, Walther C, Schoene N, Schuler G. Effects of exercise training on left ventricular function and peripheral resistance in patients with chronic heart failure: A randomized trial. JAMA. 2000 Jun 21;283(23):3095-101. doi: 10.1001/jama.283.23.3095. PMID 10865304
- [Background] Kiilavuori K, Toivonen L, Naveri H, Leinonen H. Reversal of autonomic derangements by physical training in chronic heart failure assessed by heart rate variability. Eur Heart J. 1995 Apr;16(4):490-5. doi: 10.1093/oxfordjournals.eurheartj.a060941. PMID 7671894
- [Background] Gielen S, Adams V, Mobius-Winkler S, Linke A, Erbs S, Yu J, Kempf W, Schubert A, Schuler G, Hambrecht R. Anti-inflammatory effects of exercise training in the skeletal muscle of patients with chronic heart failure. J Am Coll Cardiol. 2003 Sep 3;42(5):861-8. doi: 10.1016/s0735-1097(03)00848-9. PMID 12957433
- [Background] Adamopoulos S, Parissis J, Kroupis C, Georgiadis M, Karatzas D, Karavolias G, Koniavitou K, Coats AJ, Kremastinos DT. Physical training reduces peripheral markers of inflammation in patients with chronic heart failure. Eur Heart J. 2001 May;22(9):791-7. doi: 10.1053/euhj.2000.2285. PMID 11350112
- [Background] Shechter M, Matetzky S, Arad M, Feinberg MS, Freimark D. Vascular endothelial function predicts mortality risk in patients with advanced ischaemic chronic heart failure. Eur J Heart Fail. 2009 Jun;11(6):588-93. doi: 10.1093/eurjhf/hfp053. Epub 2009 Apr 30. PMID 19406838
- [Background] Conraads VM, Vanderheyden M, Paelinck B, Verstreken S, Blankoff I, Miljoen H, De Sutter J, Beckers P. The effect of endurance training on exercise capacity following cardiac resynchronization therapy in chronic heart failure patients: a pilot trial. Eur J Cardiovasc Prev Rehabil. 2007 Feb;14(1):99-106. doi: 10.1097/HJR.0b013e32801164b3. PMID 17301634
- [Background] Levy D, Kenchaiah S, Larson MG, Benjamin EJ, Kupka MJ, Ho KK, Murabito JM, Vasan RS. Long-term trends in the incidence of and survival with heart failure. N Engl J Med. 2002 Oct 31;347(18):1397-402. doi: 10.1056/NEJMoa020265. PMID 12409541
- [Background] Mehta PA, Dubrey SW, McIntyre HF, Walker DM, Hardman SM, Sutton GC, McDonagh TA, Cowie MR. Mode of death in patients with newly diagnosed heart failure in the general population. Eur J Heart Fail. 2008 Nov;10(11):1108-16. doi: 10.1016/j.ejheart.2008.09.004. Epub 2008 Oct 5. PMID 18838295
- [Background] Vardas PE, Auricchio A, Blanc JJ, Daubert JC, Drexler H, Ector H, Gasparini M, Linde C, Morgado FB, Oto A, Sutton R, Trusz-Gluza M; European Society of Cardiology; European Heart Rhythm Association. Guidelines for cardiac pacing and cardiac resynchronization therapy. The Task Force for Cardiac Pacing and Cardiac Resynchronization Therapy of the European Society of Cardiology. Developed in collaboration with the European Heart Rhythm Association. Europace. 2007 Oct;9(10):959-98. doi: 10.1093/europace/eum189. Epub 2007 Aug 28. No abstract available. PMID 17726043
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Fahs CA, Yan H, Ranadive S, Rossow LM, Agiovlasitis S, Wilund KR, Fernhall B. The effect of acute fish-oil supplementation on endothelial function and arterial stiffness following a high-fat meal. Appl Physiol Nutr Metab. 2010 Jun;35(3):294-302. doi: 10.1139/H10-020. PMID 20555373
- [Background] Kim J, Wang Z, Heymsfield SB, Baumgartner RN, Gallagher D. Total-body skeletal muscle mass: estimation by a new dual-energy X-ray absorptiometry method. Am J Clin Nutr. 2002 Aug;76(2):378-83. doi: 10.1093/ajcn/76.2.378. PMID 12145010
- [Background] Tomas MT, Santa-Clara MH, Monteiro E, Baynard T, Carnero EA, Bruno PM, Barroso E, Sardinha LB, Fernhall B. Body composition, muscle strength, functional capacity, and physical disability risk in liver transplanted familial amyloidotic polyneuropathy patients. Clin Transplant. 2011 Jul-Aug;25(4):E406-14. doi: 10.1111/j.1399-0012.2011.01436.x. Epub 2011 Mar 21. PMID 21418328
- [Background] Flotats A, Carrio I. Radionuclide noninvasive evaluation of heart failure beyond left ventricular function assessment. J Nucl Cardiol. 2009 Mar-Apr;16(2):304-15. doi: 10.1007/s12350-009-9064-2. Epub 2009 Feb 27. PMID 19247733
- [Background] Agostini D, Carrio I, Verberne HJ. How to use myocardial 123I-MIBG scintigraphy in chronic heart failure. Eur J Nucl Med Mol Imaging. 2009 Apr;36(4):555-9. doi: 10.1007/s00259-008-0976-x. No abstract available. PMID 18989666
- [Derived] Santa-Clara H, Abreu A, Melo X, Santos V, Cunha P, Oliveira M, Pinto R, Carmo MM, Fernhall B. High-intensity interval training in cardiac resynchronization therapy: a randomized control trial. Eur J Appl Physiol. 2019 Aug;119(8):1757-1767. doi: 10.1007/s00421-019-04165-y. Epub 2019 May 23. PMID 31123810
- [Derived] Abreu A, Oliveira M, Silva Cunha P, Santa Clara H, Portugal G, Goncalves Rodrigues I, Santos V, Morais L, Selas M, Soares R, Branco L, Ferreira R, Mota Carmo M; BETTER-HF investigators. Does permanent atrial fibrillation modify response to cardiac resynchronization therapy in heart failure patients? Rev Port Cardiol. 2017 Oct;36(10):687-694. doi: 10.1016/j.repc.2017.02.016. Epub 2017 Oct 12. English, Portuguese. PMID 29031455
- [Derived] Abreu A, Oliveira M, Silva Cunha P, Santa Clara H, Santos V, Portugal G, Rio P, Soares R, Moura Branco L, Alves M, Papoila AL, Ferreira R, Mota Carmo M; BETTER-HF investigators. Predictors of response to cardiac resynchronization therapy: A prospective cohort study. Rev Port Cardiol. 2017 Jun;36(6):417-425. doi: 10.1016/j.repc.2016.10.010. Epub 2017 May 27. English, Portuguese. PMID 28554585

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Training Program: The exercise sessions will be hospital-based, 3times a week for 60 minutes each, on non-consecutive days for 6 months. Selected the aerobic interval training (AIT) method for the development of cardiopulmonary system and the inclusion of resistance and sensorimotores exercises. The AIT comprises 4 interval training periods (high intensity) and 3 active pauses (moderate intensity) between interval training periods. The patient will warmup for 10 minutes at 50% to 60% of HRpeak from CPET, before walking to four 4 minutes intervals at 90 to 95% of HRpeak.
Period: Overall Study
Arm/Group | Exercise Training Program | Control
Started | 32 | 30
Completed | 22 | 28
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training Program | Control | Total
Number analyzed (Participants) | 22 | 28 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.8) | 66.7 (10.8) | 67.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Changes in a Composite Measure of Clinical Status - New York Heart Association Functional Class
Description: The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  I - Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. no shortness of breath when walking, climbing stairs etc.
  II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).
  Comfortable only at rest. IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Groups:
- Exercise Training Program: The exercise sessions will be hospital-based, 3times a week for 60 minutes each, on non-consecutive days for 6 months. Selected the aerobic interval training (AIT) method for the development of cardiopulmonary system and the inclusion of resistance and sensorimotores exercises. The AIT comprises 4 interval training periods (high intensity) and 3 active pauses (moderate intensity) between interval training periods.
  Exercise training program: The exercise sessions will be hospital-based, 3 times a week for 60 minutes each, on non-consecutive days for 6 months. Selected the aerobic interval training (AIT) method for the development of cardiopulmonary system and the inclusion of resistance and sensorimotores exercises. The AIT comprises 4 interval training periods (high intensity) and 3 active pauses (moderate intensity) between interval training periods. The patient will warmup for 10 minutes at 50% to 60% of HRpeak from CPET, before walking to four 4 minutes intervals at 90 to 95% of
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
scores on a scale | -1.52 [-1.82 to -1.23] | -1.0 [-1.34 to -0.65]

2. Primary Outcome: Changes in Cardiac Function - Left Ventricular Ejection Fraction
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: percentage of blood eject
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
percentage of blood eject | 11.86 [6.66 to 17.06] | 10.41 [4.69 to 16.12]

3. Primary Outcome: Changes in Exercise Testing Variables - Maximum Rate of Oxygen Consumption (VO2peak)
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: ml/kg/min
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
ml/kg/min | 2.18 [-0.53 to 4.80] | 0.25 [-2.59 to 3.09]

4. Secondary Outcome: Changes in Exercise Testing Variables - Heart Rate Recovery at 1st Minute (HRR1)
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: bpm
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
bpm | -2.19 [-12.73 to 8.35] | -15.46 [-29.35 to -1.58]

5. Secondary Outcome: Changes in Inflammatory Markers - Plasmatic Tumor Necrotic Factor Alpha (TNF-alpha)
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: µg/ml
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
µg/ml | -1.08 [-1.84 to -0.32] | 0.12 [-0.19 to 0.43]

6. Secondary Outcome: Changes in Inflammatory Markers - Plasmatic Brain Natriuretic Peptide (BNP)
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
pg/mL | -67.81 [-151.67 to 16.05] | -116.29 [-227.54 to -5.05]

7. Secondary Outcome: Changes in a Composite Measure of Quality of Life - HeartQoL T Score
Description: HeartQoL scale response of 0-3 (poor-better), higher scores indicate better quality of life. Maximum score: 42 (better prognosis); Minimum score:0 (poor prognosis)
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: t scores
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
t scores | 1.26 [0.84 to 1.68] | 0.94 [0.50 to 1.38]

8. Secondary Outcome: Changes in Exercise Testing Variables - Duration of Cardiopulmonary Testing (CPETduration)
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
seconds | 235.13 [83.07 to 387.18] | 24.00 [-50.42 to 98.42]

9. Secondary Outcome: Changes in 123I-MIBG Cardiac Scintigraphy - Heart-to-mediastinum Ratio (HMR) Early
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: mGy/MBq
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
mGy/MBq | -0.012 [-0.14 to 0.1] | -0.04 [-0.42 to 0.21]

10. Secondary Outcome: Changes in 123I-MIBG Cardiac Scintigraphy - Heart-to-mediastinum Ratio (HMR) Late
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: mGy/MBq
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
mGy/MBq | -0.07 [-0.19 to 0.05] | -0.02 [-0.3 to 0.23]

11. Secondary Outcome: Changes in 123I-MIBG Cardiac Scintigraphy - Wash Out (WO)
Description: washout provides information on the sympathetic drive. The in-vivo visualization of cardiac innervation is evaluated on planar anterior images, which are acquired early and 3 to 5 hours after tracer injection.
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
percent change | 3.56 [-2.46 to 9.59] | -3.34 [-48.13 to 34.16]

12. Secondary Outcome: Changes in Peripheral Artery Tonometry - Reactive Hyperemia (RHI)
Description: Reactive hyperaemia index (RHI) is a functional marker of endothelial dysfunction. The RHI was measured using an EndoPAT recorder.
Time Frame: 6 months after CRT implantation
Measure: Median (Inter-Quartile Range); unit: ratio of the post-to pre occlusion
Arm/Group | Exercise Training Program | Control
Number analyzed (Participants) | 22 | 28
ratio of the post-to pre occlusion | 1.1 [-1.22 to 3.34] | 0.20 [-0.17 to 0.57]

ADVERSE EVENTS:
Arm/Group | Exercise Training Program | Control
Serious Adverse Events (participants affected / at risk) | 2/22 | 3/28
Other Adverse Events (participants affected / at risk) | 0/22 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise Training Program (N=22) | Control (N=28)
Ventricular Tachycardia (Cardiac disorders) | 2 | 2
Hospital Admission (Cardiac disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No